CLINICAL TRIAL: NCT02781740
Title: Effects of Suboptimal Use of CPAP Therapy on Symptoms of Obstructive Sleep Apnoea
Brief Title: Effects of Suboptimal CPAP Therapy on Symptoms of Obstructive Sleep Apnoea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KEK-ZH-Nr.: 2016-00332; 2015-MD-0037 (Other: Swissmedic); CIV-15-12-014246 (Other: EUDAMED)
Record Dates: First submitted 2016-05-11; First posted 2016-05-24 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continous Positive Airway Pressure; CPAP; Sham CPAP; CPAP withdrawal; suboptimal CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP therapy (Active Comparator): Continuation of the already established CPAP therapy.
  Interventions: Device: Continous Positive Air Pressure Device
- Sham CPAP therapy (Sham Comparator): Sham-CPAP is achieved by setting the CPAP machine to the lowest pressure, insertion of a flow-restricting connector at the machine outlet, and insertion of six extra holes in the collar of the main tubing at the end of the mask to allow air escape and to prevent rebreathing of CO2.
  Interventions: Device: Continous Positive Air Pressure Device

INTERVENTIONS:
Device: Continous Positive Air Pressure Device

SUMMARY:
Obstructive sleep apnoea (OSA) is a highly prevalent sleep-related breathing disorder. The most effective treatment for OSA is continuous positive airway pressure (CPAP). CPAP therapy has been shown to significantly reduce subjective sleepiness and blood pressure in patients with symptomatic OSA. Its effectiveness tends to depend on its nightly usage and a commonly held view is that CPAP should be used for at least 4h/night. However, previous studies have estimated that a considerable proportion of CPAP users fail to achieve this. In addition, there is inadequate evidence to support this apparent threshold effect and so it is unclear whether such patients actually benefit from treatment or whether they could be withdrawn from CPAP, thus substantially reducing health care costs, or encouraged to increase their nightly usage of CPAP.

The aim of the proposed project is to study the effect of CPAP withdrawal on subjective sleepiness in OSA patients using CPAP for less than 4h/night on average. We hypothesize that two-week CPAP withdrawal in patients with 3-4h/night use will lead to a return of OSA-related symptoms. This trial will better establish the minimum level of CPAP adherence which could generally be regarded as effective in reducing OSA-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Objectively confirmed OSA (at the time of original diagnosis) with an oxygen desaturation index (ODI, ≥4% dips) of ≥15/h and an ESS of >10.
* Currently ≥15/h oxygen desaturations (≥4% dips) during an ambulatory nocturnal pulse oximetry performed at the end of a 4-night period without CPAP.
* Eligible patients must have been treated with CPAP for more than 12 months with a mean compliance between 3 and 4h/night. Apnoea-hypopnoea index (AHI) must be less than 10 with treatment (according to CPAP machine download data).

Exclusion Criteria:

* Previous ventilatory failure (awake PaO2<9.0kPa or arterial PaCO2>6kPa).
* Unstable, untreated coronary or peripheral artery disease, severe arterial hypertension (>180/110mmHg).
* Previously diagnosed with Cheyne-Stokes breathing.
* Current professional driver.
* Age < 20 or > 75 years at trial entry.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | Change from baseline in ESS after 2 weeks of CPAP or sham-CPAP respectively.
  Standard, well-established Epworth questionnaire. Score values between 0 and 24 represent severity of daytime sleepiness.

SECONDARY OUTCOMES:
Apnoea-Hypopnoea Index (AHI) | Change from baseline in AHI after 2 weeks of CPAP or sham-CPAP respectively.
  AHI acquired non-invasively by respiratory polygraphy at baseline and after 2 weeks. Measured in events per hour it represents severity of sleep apnoea.
Oxygen Desaturation Index (ODI) | Change from baseline in ODI after 2 weeks of CPAP or sham-CPAP respectively.
  ODI acquired non-invasively by respiratory polygraphy at baseline and after 2 weeks. Measured in events per hour it represents severity of sleep apnoea.
Mean CPAP usage time | Measured at baseline and after 2 weeks of CPAP or sham-CPAP respectively.
  Acquired automatically by the CPAP/sham-CPAP devices over the course of 2 weeks. Measured in hours per night it represents treatment adherence.
Heart rate | Change from baseline in heart rate after 2 weeks of CPAP or sham-CPAP respectively.
  Resting heart rate acquired non-invasively during wakefulness following respiratory polygraphies at baseline and after 2 weeks. Measured in beats per minute (bpm).
Mean blood pressure | Change from baseline in mean blood pressure after 2 weeks of CPAP or sham-CPAP respectively.
  Mean resting blood pressure acquired non-invasively during wakefulness following respiratory polygraphies at baseline and after 2 weeks. Measured in mmHg.
Fatigue Severity Scale (FSS) | Change from baseline in FSS after 2 weeks of CPAP or sham-CPAP respectively.
  Standard, well-established FSS questionnaire. Score values between 7 and 63 represent severity of daytime fatigue.
Quality of life as assessed in Short Form 36 (SF-36) | Change from baseline in SF-36 after 2 weeks of CPAP or sham-CPAP respectively.
  Standard, well-established 36-item patient-reported survey of patient general health status.
Quality of life as assessed in Functional Outcomes of Sleep Questionnaire 10 (FOSQ-10) | Change from baseline in FOSQ-10 after 2 weeks of CPAP or sham-CPAP respectively.
  FOSQ-10 is a standard, well-established 10-item patient-reported survey of impact of disorders of excessive sleepiness on activities of daily living.
Psychomotor vigilance as measured through the Oxford Sleep Resistance test (OSLER). | Change from baseline in OSLER after 2 weeks of CPAP or sham-CPAP respectively.
  OSLER is a standard test consisting of one to three 40-min sessions assessing the patients ability of performing a repetitive task. The OSLER error index measured in events per hour correlates statistically with sleep latency.
Psychomotor vigilance as measured through the Multiple Unprepared Reaction Time Test (MURT) | Change from baseline in MURT after 2 weeks of CPAP or sham-CPAP respectively.
  MURT is a standard test consisting of two 10-min sessions assessing the patient's alertness. The MURT time measured in milliseconds represents the patients reaction time and correlates with sleep latency.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof. Dr. med., Principal Investigator — University of Zurich
Locations (1):
- Pulmonary Division, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Gaisl T, Rejmer P, Thiel S, Haile SR, Osswald M, Roos M, Bloch KE, Stradling JR, Kohler M. Effects of suboptimal adherence of CPAP therapy on symptoms of obstructive sleep apnoea: a randomised, double-blind, controlled trial. Eur Respir J. 2020 Mar 20;55(3):1901526. doi: 10.1183/13993003.01526-2019. Print 2020 Mar. PMID 31862764